CLINICAL TRIAL: NCT02627599
Title: A Study to Evaluate Improvement in the Quality of Life and Health and Economic Outcomes of Patients Diagnosed With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Prospective Observational Study of the Breath Responsive Variable Bolus Oxygen Conserving Device
Acronym: BRVB-OCD
Status: Completed | Type: Observational
Sponsor: StratiHealth (Industry)
Collaborators: Kaiser Permanente (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 01012015DM
Record Dates: First submitted 2015-11-24; First posted 2015-12-11 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: COPD
Keywords: COPD; LTOT; Long-Term Oxygen Therapy; Oxygen Conserving Device; Quality of Life; Six Minute Walk Distance; Portable Oxygen Source; Oxygen Saturation; Breath Responsive Variable Bolus Oxygen Conserving Device; BRVB-OCD; Pulse Oximetry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic Obstructive Pulmonary Disease: * More than 12 million adults are diagnosed with COPD
  * COPD is the 3rd leading cause of death in the U.S.
  * Breathing difficulty is the major reason patients seek medical attention
  * COPD patients requiring hospitalization are associated with higher costs
  * Oximetry is an important tool for assessing need for Long-Term Oxygen Therapy
  * LTOT has been proven to improve survival and quality of life
  * Patients provided with a breath responsive variable bolus oxygen conserving device:
    1. support increased activity
    2. improve quality of life
    3. increase functional capability
    4. reduce portable oxygen source utilization
    5. maintain and/or improve oxygen saturation
  Interventions: Device: Breath Responsive Variable Bolus Oxygen Conserving Device

INTERVENTIONS:
Device: Breath Responsive Variable Bolus Oxygen Conserving Device — Mini Electronic Oxygen Conserving Device
  Other Names: SmartDose®

SUMMARY:
* Evaluate subjects in an prospective observational study
* Subjects will be administered scientifically validated questionnaires
* Evaluate Quality Improvement and Oxygen Utilization Improvements.

  1. Functional capability, dyspnea, oxygen saturation as primary endpoints
  1. Baseline Dyspnea Index (BDI)
  2. Transitional Dyspnea Index (TDI)
  3. Chronic Respiratory Disease Questionnaire (CRQ)
  4. Six minute walk distance (6MWD)
  5. Oxygen saturation using pulse oximeter
* The secondary endpoints:

  1. Portable oxygen source utilization
  2. Health care utilization (emergency room encounters, hospital admissions)

DETAILED DESCRIPTION:
Evaluate subjects in an prospective observational study in which subjects will be screened and administered scientifically validated questionnaires at study entry and during the observation period at specified intervals to determine Quality Improvements through using the Breath Responsive Variable Bolus Oxygen Conserving Device with a Portable/Ambulatory Oxygen Source on improvements in functional capability, dyspnea, oxygen saturation, quality of life as primary endpoints, and portable oxygen source utilization, health care utilization as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of chronic obstructive pulmonary disease (COPD)
* Clinically stable disease at the time of consent
* Current prescription of oxygen 24 hours a day
* Previous or current oximetry desaturation at rest or activity (≤88% on one occasion)
* Highest measured FEV1, 70% predicted; and
* Highest measured FEV1/FVC, 70% predicted
* Capable of giving informed consent
* Currently using a portable oxygen source that is a portable tank
* Mobility without a walker, cane or rollator
* Spo2 ≥ 90% on portable oxygen source at rest and activity
* Non-smoker at time of consent

Exclusion Criteria:

* Cardiovascular disease - New York Heart Association Functional Class III
* Degenerative bone or joint disease with limited functional ability
* Current homeless persons
* Active drug/alcohol dependence
* Recent drug or alcohol abuse history within the past two years
* Clinically unstable at the time of consent
* Currently a tobacco smoker

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Chronic Obstructive Pulmonary Disease
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Baseline Dyspnea Index (BDI) | At baseline once upon entry into the study
  Baseline Functional Capability, Dyspnea as measured with the Baseline Dyspnea Index (BDI)
Transition Dyspnea Index (TDI) | Every two weeks after baseline up to three months
  Improvement in Functional Capability, Dyspnea as measured with the Transition Dyspnea Index (TDI)
Chronic Respiratory Disease Questionnaire (CRQ) | At baseline upon study entry and change from baseline every two weeks up to three months
  Improvement in Quality of Life as measured with the Chronic Respiratory Disease Questionnaire
Oxygen Saturation | At baseline upon study entry and change from baseline every two weeks up to three months
  Assess pulse oximetry saturation at baseline on setting to maintain oxygen saturation equal to or greater than 90% at rest and with activity every two weeks to determine improvement or equivalence
Six Minute Walk Distance | At baseline upon study entry and change from baseline every two weeks up to three months
  Assess distance covered in meters at baseline over 6 minutes and every two weeks up to three months to determine improvement in functional capability

SECONDARY OUTCOMES:
Portable Oxygen Source Utilization | 6 Months
  Reduction in Portable Oxygen Source Use from baseline on enrollment with assessments of use each day throughout study period to determine if there are utilization reductions resulting in cost savings during study period.
Healthcare Utilization | 6 Months
  Unscheduled Hospital, Emergency Room or Physician Office Visits, as measured from baseline 6 months prior to study entry and during study period to identify utilization changes if any.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Pereira, MD, Principal Investigator — StratiHealth
Locations (3):
- United States (3):
  - KP Oceanside Medical Office Building, Oceanside, California
  - Tcmc - Mob, Vista, California
  - Pathway Medical Group, Westminster, California

IPD SHARING:
Plan to Share IPD: No
Results will be submitted for publication in peer review

REFERENCES:
- [Background] Gould GA, Scott W, Hayhurst MD, Flenley DC. Technical and clinical assessment of oxygen concentrators. Thorax. 1985 Nov;40(11):811-6. doi: 10.1136/thx.40.11.811. PMID 4071456
- [Background] Domingo C, Roig J, Coll R, Klamburg J, Izquierdo J, Ruiz-Manzano J, Morera J, Domingo E. Evaluation of the use of three different devices for nocturnal oxygen therapy in COPD patients. Respiration. 1996;63(4):230-5. doi: 10.1159/000196550. PMID 8815970
- [Background] NAUGHTON J, SEVELIUS G, BALKE B. PHYSIOLOGICAL RESPONSES OF NORMAL AND PATHOLOGICAL SUBJECTS TO A MODIFIED WORK CAPACITY TEST. J Sports Med Phys Fitness. 1963 Dec;3:201-7. No abstract available. PMID 14099069
- [Background] Hankinson JL, Odencrantz JR, Fedan KB. Spirometric reference values from a sample of the general U.S. population. Am J Respir Crit Care Med. 1999 Jan;159(1):179-87. doi: 10.1164/ajrccm.159.1.9712108. PMID 9872837
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Carter R, Tashkin D, Djahed B, Hathaway E, Nicotra MB, Tiep BL. Demand oxygen delivery for patients with restrictive lung disease. Chest. 1989 Dec;96(6):1307-11. doi: 10.1378/chest.96.6.1307. PMID 2582836
- [Background] Rinow ME, Saltzman AR. Effectiveness of a new oxygen demand valve in chronic hypoxemia. Chest. 1986 Aug;90(2):204-7. doi: 10.1378/chest.90.2.204. PMID 3731892
- [Background] Tiep BL, Nicotra MB, Carter R, Phillips R, Otsap B. Low-concentration oxygen therapy via a demand oxygen delivery system. Chest. 1985 May;87(5):636-8. doi: 10.1378/chest.87.5.636. PMID 3921316
- [Background] Moore-Gillon JC, George RJ, Geddes DM. An oxygen conserving nasal cannula. Thorax. 1985 Nov;40(11):817-9. doi: 10.1136/thx.40.11.817. PMID 4071457
- [Result] Cranston JM, Crockett AJ, Moss JR, Alpers JH. Domiciliary oxygen for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2005 Oct 19;2005(4):CD001744. doi: 10.1002/14651858.CD001744.pub2. PMID 16235285
- [Result] Celli BR, MacNee W; ATS/ERS Task Force. Standards for the diagnosis and treatment of patients with COPD: a summary of the ATS/ERS position paper. Eur Respir J. 2004 Jun;23(6):932-46. doi: 10.1183/09031936.04.00014304. No abstract available. PMID 15219010
- [Result] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Result] Strickland SL, Hogan TM, Hogan RG, Sohal HS, McKenzie WN, Petroski GF. A randomized multi-arm repeated-measures prospective study of several modalities of portable oxygen delivery during assessment of functional exercise capacity. Respir Care. 2009 Mar;54(3):344-9. PMID 19245728
- [Result] Fuhrman C, Chouaid C, Herigault R, Housset B, Adnot S. Comparison of four demand oxygen delivery systems at rest and during exercise for chronic obstructive pulmonary disease. Respir Med. 2004 Oct;98(10):938-44. doi: 10.1016/j.rmed.2004.03.010. PMID 15481269
- [Result] Langenhof S, Fichter J. Comparison of two demand oxygen delivery devices for administration of oxygen in COPD. Chest. 2005 Oct;128(4):2082-7. doi: 10.1378/chest.128.4.2082. PMID 16236858
- [Result] Garrod R, Bestall JC, Paul E, Wedzicha JA. Evaluation of pulsed dose oxygen delivery during exercise in patients with severe chronic obstructive pulmonary disease. Thorax. 1999 Mar;54(3):242-4. doi: 10.1136/thx.54.3.242. PMID 10325901
- [Result] Gallegos LC, Shigeoka JW. Novel oxygen-concentrator-based equipment: take a test drive first! Respir Care. 2006 Jan;51(1):25-8. No abstract available. PMID 16381613
- [Result] Jette M, Sidney K, Blumchen G. Metabolic equivalents (METS) in exercise testing, exercise prescription, and evaluation of functional capacity. Clin Cardiol. 1990 Aug;13(8):555-65. doi: 10.1002/clc.4960130809. PMID 2204507
- [Result] Bliss PL, McCoy RW, Adams AB. Characteristics of demand oxygen delivery systems: maximum output and setting recommendations. Respir Care. 2004 Feb;49(2):160-5. PMID 14744265
- [Result] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Result] Palwai A, Skowronski M, Coreno A, Drummond C, McFadden ER Jr. Critical comparisons of the clinical performance of oxygen-conserving devices. Am J Respir Crit Care Med. 2010 May 15;181(10):1061-71. doi: 10.1164/rccm.200910-1638OC. Epub 2010 Feb 4. PMID 20133925
- [Result] Senn S, Wanger J, Fernandez E, Cherniack RM. Efficacy of a pulsed oxygen delivery device during exercise in patients with chronic respiratory disease. Chest. 1989 Sep;96(3):467-72. doi: 10.1378/chest.96.3.467. PMID 2766806
- [Result] Bower JS, Brook CJ, Zimmer K, Davis D. Performance of a demand oxygen saver system during rest, exercise, and sleep in hypoxemic patients. Chest. 1988 Jul;94(1):77-80. doi: 10.1378/chest.94.1.77. PMID 3383659
- [Result] Tiep BL, Carter R, Nicotra B, Berry J, Phillips RE, Otsap B. Demand oxygen delivery during exercise. Chest. 1987 Jan;91(1):15-20. doi: 10.1378/chest.91.1.15. PMID 3792073
- [Result] Mecikalski M, Shigeoka JW. A demand valve conserves oxygen in subjects with chronic obstructive pulmonary disease. Chest. 1984 Nov;86(5):667-70. doi: 10.1378/chest.86.5.667. PMID 6488901
- [Result] Roberts CM, Bell J, Wedzicha JA. Comparison of the efficacy of a demand oxygen delivery system with continuous low flow oxygen in subjects with stable COPD and severe oxygen desaturation on walking. Thorax. 1996 Aug;51(8):831-4. doi: 10.1136/thx.51.8.831. PMID 8795673
- [Result] Braun SR, Spratt G, Scott GC, Ellersieck M. Comparison of six oxygen delivery systems for COPD patients at rest and during exercise. Chest. 1992 Sep;102(3):694-8. doi: 10.1378/chest.102.3.694. PMID 1516389
- [Result] McCoy R. Oxygen-conserving techniques and devices. Respir Care. 2000 Jan;45(1):95-103; discussion 104. PMID 10771785
- [Result] Doherty DE, Petty TL, Bailey W, Carlin B, Cassaburi R, Christopher K, Kvale P, Make B, Mapel D, Selecky P, Tiger J. Recommendations of the 6th long-term oxygen therapy consensus conference. Respir Care. 2006 May;51(5):519-25. No abstract available. PMID 16710952
- [Result] Long term domiciliary oxygen therapy in chronic hypoxic cor pulmonale complicating chronic bronchitis and emphysema. Report of the Medical Research Council Working Party. Lancet. 1981 Mar 28;1(8222):681-6. PMID 6110912
- [Result] Continuous or nocturnal oxygen therapy in hypoxemic chronic obstructive lung disease: a clinical trial. Nocturnal Oxygen Therapy Trial Group. Ann Intern Med. 1980 Sep;93(3):391-8. doi: 10.7326/0003-4819-93-3-391. PMID 6776858
- [Result] Hardinge M, Annandale J, Bourne S, Cooper B, Evans A, Freeman D, Green A, Hippolyte S, Knowles V, MacNee W, McDonnell L, Pye K, Suntharalingam J, Vora V, Wilkinson T; British Thoracic Society Home Oxygen Guideline Development Group; British Thoracic Society Standards of Care Committee. British Thoracic Society guidelines for home oxygen use in adults. Thorax. 2015 Jun;70 Suppl 1:i1-43. doi: 10.1136/thoraxjnl-2015-206865. PMID 25870317
- [Result] Marti S, Pajares V, Morante F, Ramon MA, Lara J, Ferrer J, Guell MR. Are oxygen-conserving devices effective for correcting exercise hypoxemia? Respir Care. 2013 Oct;58(10):1606-13. doi: 10.4187/respcare.02260. Epub 2013 Mar 19. PMID 23513249
- [Result] Petty TL, Bliss PL. Ambulatory oxygen therapy, exercise, and survival with advanced chronic obstructive pulmonary disease (the Nocturnal Oxygen Therapy Trial revisited). Respir Care. 2000 Feb;45(2):204-11; discussion 211-3. PMID 10771792
- [Result] Tiep BL, Lewis MI. Oxygen conservation and oxygen-conserving devices in chronic lung disease. A review. Chest. 1987 Aug;92(2):263-72. doi: 10.1378/chest.92.2.263. PMID 3608597
- [Result] Pertelle, VR, Oxygen Conserving Technologies: Device Variability and the Effect on Clinical Applications and Expected Outcomes: A White Paper, October 2015